CLINICAL TRIAL: NCT01861639
Title: Effect of Repetitive Transcranial Magnetic Stimulation (rTMS) on Cognition and Brain Networks in Healthy Subjects in 2 Sessions 15 Days Apart
Brief Title: Stability of rTMS on Cognition and Brain Networks on Healthy Subjects.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Timeframe of the IMI project couldn't be expended
Sponsor: Qualissima (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: WP1P003
Record Dates: First submitted 2013-05-16; First posted 2013-05-23 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
MeSH Terms: interventions — Magnetic Resonance Imaging; Electroencephalography

STUDY DESIGN:
Who Masked: Participant

ARMS (8):
- ineffective rTMS - Active TBS - fMRI (Experimental)
  Interventions: Device: ineffective rTMS; Device: active TBS; Device: fMRI
- Effective rTMS - Active TBS - fMRI (Experimental)
  Interventions: Device: active TBS; Device: fMRI; Device: Effective rTMS
- ineffective rTMS - Sham TBS - fMRI (Sham Comparator)
  Interventions: Device: ineffective rTMS; Device: Sham TBS; Device: fMRI
- Effective rTMS - Sham TBS - fMRI (Sham Comparator)
  Interventions: Device: Sham TBS; Device: fMRI; Device: Effective rTMS
- ineffective rTMS - Active TBS - EEG (Experimental)
  Interventions: Device: ineffective rTMS; Device: active TBS; Device: EEG
- Effective rTMS - Active TBS - EEG (Experimental)
  Interventions: Device: active TBS; Device: EEG; Device: Effective rTMS
- ineffective rTMS - Sham TBS - EEG (Sham Comparator)
  Interventions: Device: ineffective rTMS; Device: Sham TBS; Device: EEG
- Effective rTMS - Sham TBS - EEG (Sham Comparator)
  Interventions: Device: Sham TBS; Device: EEG; Device: Effective rTMS

INTERVENTIONS:
Device: ineffective rTMS — A 20Hz repetitive transcranial magnetic stimulation (rTMS) will be applied for 900 ms with an intensity of 90% of motor threshold. Active stimulation will be applied on the L-DLPFC compared to an ineffective stimulation.
  Arms: ineffective rTMS - Active TBS - EEG; ineffective rTMS - Active TBS - fMRI; ineffective rTMS - Sham TBS - EEG; ineffective rTMS - Sham TBS - fMRI
Device: active TBS — A continuous Theta-Burst Stimulation (cTBS) protocol will be applied over the L-DLPFC. Three stimuli at 50Hz, 80% of individual Motor Threshold will be repeated every 200ms for 40sec
  Arms: Effective rTMS - Active TBS - EEG; Effective rTMS - Active TBS - fMRI; ineffective rTMS - Active TBS - EEG; ineffective rTMS - Active TBS - fMRI
Device: Sham TBS — A Sham stimulation will be applied over the L-DLPFC. a placebo coil will be used.
  Arms: Effective rTMS - Sham TBS - EEG; Effective rTMS - Sham TBS - fMRI; ineffective rTMS - Sham TBS - EEG; ineffective rTMS - Sham TBS - fMRI
Device: fMRI — Functional MRI data will be acquired during the performance of the memory task. Functional data will be acquired with a blood oxygenation level dependant (BOLD) contrast sensitive gradient echo, T2*-weighted echo-planar imaging sequence
  Arms: Effective rTMS - Active TBS - fMRI; Effective rTMS - Sham TBS - fMRI; ineffective rTMS - Active TBS - fMRI; ineffective rTMS - Sham TBS - fMRI
Device: EEG — EEG will be coupled with task performance in an event-related manner to be able to isolate brain activity of each type of stimuli presented. EEG imaging data will be acquired during the memory task.
  Arms: Effective rTMS - Active TBS - EEG; Effective rTMS - Sham TBS - EEG; ineffective rTMS - Active TBS - EEG; ineffective rTMS - Sham TBS - EEG
Device: Effective rTMS — A 20Hz repetitive transcranial magnetic stimulation (rTMS) will be applied for 900 ms with an intensity of 90% of motor threshold. Active stimulation will be applied on the L-DLPFC compared to an effective stimulation.
  Arms: Effective rTMS - Active TBS - EEG; Effective rTMS - Active TBS - fMRI; Effective rTMS - Sham TBS - EEG; Effective rTMS - Sham TBS - fMRI

SUMMARY:
Episodic and working memory processes are the most affected cognitive domains in Alzheimer's Disease (AD) and its early stage, Mild Cognitive Impairment (MCI).

Transcranial Magnetic Stimulation (TMS) is a unique tool to interfere with cognitive processes by inducing "virtual and transient lesions", mimicking those observed in MCI. It has proven repeatedly its capacity to interfere with encoding-retrieval memory task. However, to date, only few imaging data exist on the cerebral pathways involved in encoding memory task. Moreover, the stability of TMS effects over time remains to be investigated. If proven to be a stable interfering challenge, TMS could be used to investigate the potential restoring effect of new medication in AD.

The study is the pilot study of a larger clinical trial which aims to prove the utility of rTMS as a potential model for prediction of clinical efficacy using a combination of cognitive and neuroimaging endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged between 18 and 40 years-old inclusive.
* Education level: at least secondary.
* Right-handed (Edinburgh Handedness Inventory).
* The subjects are in good health on the basis of the medical interview (medical history, symptoms), the physical examination and vital signs.
* No history of psychiatric disorders (assessed by Structured Clinical Interview for DSM IV Disorders (SCID) for Barcelona and by the Mini International Neuropsychiatric Interview (MINI) for Marseille).
* No history of neurological disorders
* No history of concussion (cranial or facial trauma) without or with loss of consciousness.
* Subject without history of brain disease (severe brain trauma, stroke, cerebral tumor...).
* Subject without lesion on MRI.
* Subject without abnormal electrical activities on standard clinical EEG.
* No history of drug or alcohol abuse.
* No smoker or ≤ 5 cg/ day.
* The subject can complete the neuropsychological test battery during the training session.
* Subject without contraindication to MRI.
* The subject is able to read and understand the Information Form and comply with the protocol instructions and restrictions.
* The subject is covered by a social insurance.
* The subject has provided written informed consent.

Exclusion Criteria:

* History or presence of psychiatric illness (Psychiatric interview).
* History or presence of neurologic illness.
* The subject, in the opinion of the investigator, is unlikely to comply with the study protocol or is unsuitable for any other reason.
* The subject participates in another clinical trial or is still being within a washout period of 1 month since last taking of a previous clinical trial, or subjects who have received more than 4500 Euros in the previous 12 months for participating in clinical trials.
* Presence of metallic objects within the body.
* Subjects with pacemaker.
* Claustrophobia.
* Individual and familial history of epileptic seizure.
* Any medication listed (see annexe) in the safety guidelines published by the Safety of TMS Consensus Group (Rossi et al., 2009) will be forbidden.
* Subject with a correct hit rate during the retrieval session of the memory task

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2013-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Outputs of the memory task | up to Day 15
  outputs: number of correct answers during the retrieval event-related task (Hit rate) and the rate of false recognition of novel pictures (False Alarms rate).

SECONDARY OUTCOMES:
CANTAB task | Day 1 and Day 15
  * CANTAB / Rapid Visual Information Processing (RVIP)
  * CANTAB / Spatial Working Memory (SWM)
  * CANTAB / Paired Associates Learning (PAL)
Gene expression | Day 1
  Interest genes expression will be investigated depending on the impact of TMS on behavioral and functional brain responses.
Imaging | Day1 and Day 15
  Functional MRI (Barcelona): modifications will be highlighted by changes in Blood Oxydation level Dependence (BOLD)signal patterns
  EEG (Marseille): modifications will be highlighted by changes in EEG markers

CONTACTS AND LOCATIONS:
Overall Officials: David Bartrés-Faz, Principal Investigator — Institut d'Investigacions Biomèdiques August Pi i Sunyer; Christine Audebert, Principal Investigator — CIC-CPCET
Locations (2):
- Cic-Cpcet, Marseille, France
- IDIBAPS, Barcelona, Spain